CLINICAL TRIAL: NCT03493542
Title: A Phase 3 Open-Label Clinical Trial to Study the Immunogenicity, Safety and Tolerability of Recombinant Human Papillomavirus Quadrivalent (Types 6, 11, 16, 18) Vaccine (V501) in Chinese Girls Aged 9-19 Years and Young Women Aged 20-26 Years
Brief Title: A Study to Evaluate the Immunogenicity, Safety and Tolerability of Quadrivalent Human Papillomavirus Vaccine (V501) in Chinese Girls Aged 9-19 Years and Young Women Aged 20-26 Years (V501-213)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V501-213; V501-213 (Other: MSD Protocol Number); 2023-001144-29 (EudraCT Number)
Record Dates: First submitted 2018-04-04; First posted 2018-04-10 (Actual); Results first posted 2020-05-04 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Prevention of HPV Types 16- and 18-related Cervical Cancer, Cervical Intraepithelial Neoplasia (CIN) 1/2/3, and Cervical Adenocarcinoma in Situ
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; Vaccines, Synthetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Chinese Girls Aged 9 to 19 Years (Experimental): Participants will receive V501 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6
  Interventions: Biological: V501
- Chinese Young Women Aged 20 to 26 Years (Active Comparator): Participants will receive V501 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6
  Interventions: Biological: V501

INTERVENTIONS:
Biological: V501 — 0.5 mL intramuscular injection in the deltoid muscle at Day 1, Month 2, and Month 6
  Other Names: (Gardasil®) human papillomavirus (types 6, 11, 16, 18) recombinant vaccine; qHPV

SUMMARY:
This study is designed to evaluate the immunogenicity, safety, and tolerability of Gardasil® (quadrivalent human papillomavirus [qHPV] vaccine, V501) in Chinese girls aged 9-19 years and young women aged 20-26 years. The primary hypothesis of the study states that at 1 month postdose 3, a 3-dose regimen of V501 induces non-inferior geometric mean titers (GMTs) for serum anti-HPV 6, anti-HPV 11, anti-HPV 16, anti-HPV 18 in girls aged 9-19 years compared to young women aged 20-26 years.

DETAILED DESCRIPTION:
The study consists of a Base Stage wherein Chinese girls aged 9-19 years and young women aged 20-26 years receive a 3-dose regimen of V501 and are followed up to 1 month postdose 3 (Month 7). Participants aged 9-19 years who received 3 doses of V501 in the Base Stage will be eligible to participate in the Extension Stage and will be followed up to Month 60. No study vaccine will be administered during the Extension Stage.

ELIGIBILITY:
Inclusion Criteria:

* Not pregnant and 1) not a woman of childbearing potential (WOCBP), or 2) a WOCBP who has not had sex with males or has had sex with males and used effective contraception since the first day of participant's last menstrual period through Day 1 and understands and agrees that during the study she should not have sexual intercourse with males without effective contraception (the rhythm method, withdrawal, and emergency contraception are not acceptable methods per the protocol).
* Participant and participant's parent or guardian (participants aged 9-17 years only) provided written informed consent/assent.
* Provided a primary and alternative telephone for follow-up purposes.
* Extension Stage: participant was enrolled in the 9-19 years old group, received 3 doses of V501 in the Base Stage, and participant and participant's legally acceptable representative (if applicable) provided written informed consent/assent for the study extension.

Exclusion Criteria:

* History of severe allergic reaction that required medical intervention.
* Allergic to any vaccine component, including aluminum, yeast, or Benzonase® (nuclease).
* Known thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injections.
* Currently immunocompromised or was diagnosed as having congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammatory bowel disease, or other autoimmune condition.
* History of splenectomy.
* Any condition which in the opinion of the investigator might interfere with the evaluation of the study objectives.
* History of recent or ongoing alcohol or other drug abuse.
* History of a positive test for HPV.
* Any history of abnormal Pap test.
* History of external genital wart, vulvar intraepithelial neoplasia (VIN), vaginal intraepithelial neoplasia (VaIN), vulvar cancer or vaginal cancer.
* Undergone hysterectomy (either vaginal or total abdominal hysterectomy).
* Receiving or has received in the year prior to Day 1 vaccination an excluded immunosuppressive therapy. A participant will be excluded if she is currently receiving steroid therapy, has recently received such therapy, or has received 2 or more courses of corticosteroids (orally or parenterally) lasting at least 1 week in duration in the year prior to Day 1 vaccination. Participants using inhaled, nasal or topical steroids are considered eligible for the study.
* Received immune globulin product or blood-derived product within 6 months prior to Day 1 vaccination, or plans to receive any such product during the study.
* Received a marketed HPV vaccine, or has participated in an HPV vaccine clinical trial and has received either active agent or placebo.
* Received inactivated or recombinant vaccines within 14 days prior to Day 1 vaccination or receipt of live vaccines within 21 days prior to Day 1 vaccination.
* Concurrently enrolled in a clinical study of investigational agents.
* Had >4 lifetime sexual partners.
* Unlikely to adhere to the study procedures, keep appointments, or is planning to permanently relocate from the area prior to the completion of the study or to leave for an extended period of time when study visits would need to be scheduled.
* An immediate family member who is investigational site or sponsor staff directly involved with this study.
* Extension Stage: reported overdose or received non-study HPV vaccine during the Base Stage.

Ages: 9 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 766 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Yangchun Center For Disease Prevention And Control ( Site 0003), Yangchun, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Huang Z, He J, Su J, Ou Z, Liu G, Fu R, Shou Q, Zheng M, Group T, Luxembourg A, Liao X, Zhang J. Immunogenicity and safety of the quadrivalent human papillomavirus vaccine in Chinese females aged 9 to 26 years: A phase 3, open-label, immunobridging study. Vaccine. 2021 Jan 22;39(4):760-766. doi: 10.1016/j.vaccine.2020.11.008. Epub 2020 Nov 22. PMID 33239228
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Base Study: Chinese Girls Aged 9 to 19 Years; Base Study: Chinese Young Women Aged 20 to 26 Years: Participants received V501 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6
- Extension Study: Chinese Girls Aged 9 to 19 Years: In base study, participants received V501 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6 and followed up to Month 7. In the extension studies after Month 7, the participants were followed up for safety and immunogenicity up to Month 60 (EXT)
Period: Base Study
Arm/Group | Base Study: Chinese Girls Aged 9 to 19 Years | Base Study: Chinese Young Women Aged 20 to 26 Years | Extension Study: Chinese Girls Aged 9 to 19 Years
Started | 383 | 383 | 0
Vaccination 1 | 383 | 383 | 0
Vaccination 2 | 379 | 378 | 0
Vaccination 3 | 378 | 377 | 0
Completed | 383 | 379 | 0
Not Completed | 0 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 0
Period: Extension Study
Arm/Group | Base Study: Chinese Girls Aged 9 to 19 Years | Base Study: Chinese Young Women Aged 20 to 26 Years | Extension Study: Chinese Girls Aged 9 to 19 Years
Started | 0 | 0 | 365
Completed | 0 | 0 | 338
Not Completed | 0 | 0 | 27
Not completed — Consent withdrawal by parent/guardian | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 25

BASELINE CHARACTERISTICS:
Population: Per protocol, baseline characteristics were analyzed in all participants randomized in the base study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Base Study: Chinese Girls Aged 9 to 19 Years | Base Study: Chinese Young Women Aged 20 to 26 Years | Total
Number analyzed (Participants) | 383 | 383 | 766
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (3.3) | 23.4 (1.8) | 18.8 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 383 | 383 | 766
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 383 | 383 | 766
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 383 | 383 | 766
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Base Stage: Geometric Mean Titers for Serum Anti-Human Papillomavirus (HPV) Types 6, 11, 16, and 18: Competitive Luminex Immunoassay (cLIA)
Description: Serum antibody titers (Geometric mean titers) for HPV Types 6, 11, 16, and 18 were measured. Antibodies were measured using a Competitive Luminex Immunoassay (cLIA). Antibody titers were expressed as milli Merck Units/milliliter (mMU/mL).
Time Frame: Month 7 (1 month postdose 3)
Population: Per protocol, the analysis population included the participants with immune response to each of the 4 HPV types (6, 11, 16, and 18), who received 3 vaccinations and met following criteria: received all 3 vaccinations within acceptable day ranges, seronegative at Day 1 for HPV type(s), had a Day 1 through Month 7 serum sample collected within an acceptable day range, and had no protocol violation that potentially interfered with the evaluation of immune responses to the qHPV vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Groups:
- Chinese Girls Aged 9 to 19 Years; Base Study: Chinese Young Women Aged 20 to 26 Years: Participants received V501 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6
Arm/Group | Chinese Girls Aged 9 to 19 Years | Base Study: Chinese Young Women Aged 20 to 26 Years
Number analyzed (Participants) | 383 | 383
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 343 | 315
  Anti-HPV 6 | 975.2 [905.6 to 1050.2] | 686.6 [635.5 to 741.7]
  Anti-HPV 11: number analyzed (Participants) | 343 | 315
  Anti-HPV 11 | 807.4 [749.8 to 869.4] | 580.2 [537.0 to 626.8]
  Anti-HPV 16: number analyzed (Participants) | 354 | 330
  Anti-HPV 16 | 4573.7 [4244.5 to 4928.3] | 2989.2 [2766.7 to 3229.6]
  Anti-HPV 18: number analyzed (Participants) | 333 | 318
  Anti-HPV 18 | 1176.5 [1069.0 to 1294.8] | 708.6 [642.4 to 781.6]
Statistical Analysis 1: Comparison: Chinese Girls Aged 9 to 19 Years vs Base Study: Chinese Young Women Aged 20 to 26 Years; Anti-HPV 6; Test type: Non-Inferiority — The statistical criterion for non-inferiority required that the lower bound of two-sided 95% confidence interval of GMT ratio (9 to 19 years old/20 to 26 years old) was greater than 0.67 for each HPV type; p < 0.0001, ANOVA; GMT Ratio = 1.42, 95% CI 2-sided [1.28 to 1.58] — GMT Ratio = GMT (9-19 yr)/GMT(20-26 yr)
Statistical Analysis 2: Comparison: Chinese Girls Aged 9 to 19 Years vs Base Study: Chinese Young Women Aged 20 to 26 Years; Anti-HPV 11; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; GMT Ratio = 1.39, 95% CI 2-sided [1.25 to 1.55] — GMT Ratio = GMT (9-19 yr)/GMT(20-26 yr)
Statistical Analysis 3: Comparison: Chinese Girls Aged 9 to 19 Years vs Base Study: Chinese Young Women Aged 20 to 26 Years; Anti-HPV 16; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; GMT Ratio = 1.53, 95% CI 2-sided [1.37 to 1.70] — GMT Ratio = GMT (9-19 yr)/GMT(20-26 yr)
Statistical Analysis 4: Comparison: Chinese Girls Aged 9 to 19 Years vs Base Study: Chinese Young Women Aged 20 to 26 Years; Anti-HPV 18; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; GMT Ratio = 1.66, 95% CI 2-sided [1.45 to 1.90] — GMT Ratio = GMT (9-19 yr)/GMT(20-26 yr)

2. Primary Outcome: Extension Stage: GMTs for Serum Anti-Human Papillomavirus (HPV) Types 6, 11, 16, and 18 at Month 12 Assessed by cLIA
Description: Serum antibody titers (Geometric mean titers) for HPV Types 6, 11, 16, and 18 were measured. Antibodies were measured using a Competitive Luminex Immunoassay (cLIA). Antibody titers were expressed as (mMU/mL).
Time Frame: Month 12 post-vaccination 1
Population: Per protocol, the analysis population included participants with immune response to each of the 4 HPV types (6, 11, 16, and 18), who received 3 vaccinations and met following criteria: received all 3 vaccinations within acceptable day ranges, seronegative at Day 1 for HPV type(s), had a Day 1 through Month 7 serum sample collected within an acceptable day range, and had no protocol violation that potentially interfered with the evaluation of immune responses to the qHPV vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Years
Number analyzed (Participants) | 365
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 328
  Anti-HPV 6 | 259.1 [237.6 to 282.4]
  Anti-HPV 11: number analyzed (Participants) | 328
  Anti-HPV 11 | 206.7 [190.5 to 224.3]
  Anti-HPV 16: number analyzed (Participants) | 338
  Anti-HPV 16 | 1149.8 [1054.6 to 1253.7]
  Anti-HPV 18: number analyzed (Participants) | 320
  Anti-HPV 18 | 284.2 [257.3 to 313.8]

3. Primary Outcome: Extension Stage: GMTs for Serum Anti-Human Papillomavirus (HPV) Types 6, 11, 16, and 18 at Month 24 Assessed by cLIA
Description: as for outcome 2
Time Frame: Month 24 post-vaccination 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Years
Number analyzed (Participants) | 365
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 322
  Anti-HPV 6 | 137.9 [125.5 to 151.4]
  Anti-HPV 11: number analyzed (Participants) | 322
  Anti-HPV 11 | 110.3 [101.0 to 120.6]
  Anti-HPV 16: number analyzed (Participants) | 333
  Anti-HPV 16 | 522.6 [472.1 to 578.5]
  Anti-HPV 18: number analyzed (Participants) | 316
  Anti-HPV 18 | 157.2 [142.7 to 173.3]

4. Primary Outcome: Extension Stage: GMTs for Serum Anti-Human Papillomavirus (HPV) Types 6, 11, 16, and 18 at Month 36 Assessed by cLIA
Description: as for outcome 2
Time Frame: Month 36 post-vaccination 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Years
Number analyzed (Participants) | 365
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 318
  Anti-HPV 6 | 110.6 [101.3 to 120.7]
  Anti-HPV 11: number analyzed (Participants) | 318
  Anti-HPV 11 | 87.0 [79.6 to 95.2]
  Anti-HPV 16: number analyzed (Participants) | 329
  Anti-HPV 16 | 400.8 [359.5 to 446.8]
  Anti-HPV 18: number analyzed (Participants) | 312
  Anti-HPV 18 | 131.9 [120.2 to 144.8]

5. Primary Outcome: Extension Stage: GMTs for Serum Anti-Human Papillomavirus (HPV) Types 6, 11, 16, and 18 at Month 48 Assessed by cLIA
Description: as for outcome 2
Time Frame: Month 48 post-vaccination 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Years
Number analyzed (Participants) | 365
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 311
  Anti-HPV 6 | 103.0 [94.4 to 112.4]
  Anti-HPV 11: number analyzed (Participants) | 311
  Anti-HPV 11 | 81.8 [74.8 to 89.3]
  Anti-HPV 16: number analyzed (Participants) | 321
  Anti-HPV 16 | 347.5 [310.0 to 389.6]
  Anti-HPV 18: number analyzed (Participants) | 305
  Anti-HPV 18 | 130.3 [118.9 to 142.7]

6. Primary Outcome: Extension Stage: GMTs for Serum Anti-Human Papillomavirus (HPV) Types 6, 11, 16, and 18 at Month 60 Assessed by cLIA
Description: Serum antibody titers (Geometric mean titers) for HPV virus-like particles (VLPs) Types 6, 11, 16, and 18 were measured. Antibodies were measured using a Competitive Luminex Immunoassay (cLIA). Antibody titers were expressed as (mMU/mL).
Time Frame: Month 60 post-vaccination 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Years
Number analyzed (Participants) | 365
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 307
  Anti-HPV 6 | 87.6 [80.4 to 95.4]
  Anti-HPV 11: number analyzed (Participants) | 307
  Anti-HPV 11 | 67.3 [61.6 to 73.5]
  Anti-HPV 16: number analyzed (Participants) | 317
  Anti-HPV 16 | 283.2 [250.8 to 319.8]
  Anti-HPV 18: number analyzed (Participants) | 302
  Anti-HPV 18 | 113.6 [103.7 to 124.5]

7. Primary Outcome: Extension Stage: Percentage of Participants With Seropositivity to HPV Types 6, 11, 16, and 18 at Month 12 Assessed by cLIA
Description: The percentage of participants who are seropositive to each of HPV Types 6, 11, 16, and 18 were assessed. Antibodies were measured using cLIA.
Time Frame: Month 12 post-vaccination 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Extension Study: Chinese Girls Aged 9 to 19 Year: In base study, participants received V501 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6 and followed up to Month 7. In the extension studies after Month 7, the participants were followed up for safety and immunogenicity up to Month 60 (EXT)
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Year
Number analyzed (Participants) | 365
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 328
  Anti-HPV 6 | 99.1 [97.4 to 99.8]
  Anti-HPV 11: number analyzed (Participants) | 328
  Anti-HPV 11 | 99.7 [98.3 to 100.0]
  Anti-HPV 16: number analyzed (Participants) | 338
  Anti-HPV 16 | 100.0 [98.9 to 100.0]
  Anti-HPV 18: number analyzed (Participants) | 320
  Anti-HPV 18 | 96.9 [94.3 to 98.5]

8. Primary Outcome: Extension Stage: Percentage of Participants With Seropositivity to HPV Types 6, 11, 16, and 18 at Month 24 Assessed by cLIA
Description: as for outcome 7
Time Frame: Month 24 post-vaccination 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Year
Number analyzed (Participants) | 365
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 322
  Anti-HPV 6 | 88.8 [84.9 to 92.0]
  Anti-HPV 11: number analyzed (Participants) | 322
  Anti-HPV 11 | 95.3 [92.4 to 97.4]
  Anti-HPV 16: number analyzed (Participants) | 333
  Anti-HPV 16 | 99.7 [98.3 to 100.0]
  Anti-HPV 18: number analyzed (Participants) | 316
  Anti-HPV 18 | 87.7 [83.5 to 91.1]

9. Primary Outcome: Extension Stage: Percentage of Participants With Seropositivity to HPV Types 6, 11, 16, and 18 at Month 36 Assessed by cLIA
Description: as for outcome 7
Time Frame: Month 36 post-vaccination 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Year
Number analyzed (Participants) | 365
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 318
  Anti-HPV 6 | 83.6 [79.1 to 87.5]
  Anti-HPV 11: number analyzed (Participants) | 318
  Anti-HPV 11 | 92.1 [88.6 to 94.8]
  Anti-HPV 16: number analyzed (Participants) | 329
  Anti-HPV 16 | 98.8 [96.9 to 99.7]
  Anti-HPV 18: number analyzed (Participants) | 312
  Anti-HPV 18 | 84.0 [79.4 to 87.9]

10. Primary Outcome: Extension Stage: Percentage of Participants With Seropositivity to HPV Types 6, 11, 16, and 18 at Month 48 Assessed by cLIA
Description: as for outcome 7
Time Frame: Month 48 post-vaccination 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Year
Number analyzed (Participants) | 365
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 311
  Anti-HPV 6 | 68.5 [63.0 to 73.6]
  Anti-HPV 11: number analyzed (Participants) | 311
  Anti-HPV 11 | 85.2 [80.8 to 89.0]
  Anti-HPV 16: number analyzed (Participants) | 321
  Anti-HPV 16 | 91.9 [88.4 to 94.6]
  Anti-HPV 18: number analyzed (Participants) | 305
  Anti-HPV 18 | 64.6 [58.9 to 70.0]

11. Primary Outcome: Extension Stage: Percentage of Participants With Seropositivity to HPV Types 6, 11, 16, and 18 at Month 60 Assessed by cLIA
Description: as for outcome 7
Time Frame: Month 60 post-vaccination 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Year
Number analyzed (Participants) | 365
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 307
  Anti-HPV 6 | 61.9 [56.2 to 67.3]
  Anti-HPV 11: number analyzed (Participants) | 307
  Anti-HPV 11 | 74.9 [69.7 to 79.7]
  Anti-HPV 16: number analyzed (Participants) | 317
  Anti-HPV 16 | 87.1 [82.9 to 90.6]
  Anti-HPV 18: number analyzed (Participants) | 302
  Anti-HPV 18 | 58.3 [52.5 to 63.9]

12. Primary Outcome: Extension Stage: GMTs for Serum Anti-HPV Types 6, 11, 16, and 18 at Month 12 Assessed by Immunoglobulin G Luminex Immunoassay (IgG LIA)
Description: Serum antibody titers (Geometric mean titers) for HPV Types 6, 11, 16, and 18 were measured. Antibodies were measured using IgG LIA. Antibody titers were expressed as (mMU/mL).
Time Frame: Month 12 post-vaccination 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Years
Number analyzed (Participants) | 365
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 328
  Anti-HPV 6 | 217.0 [198.1 to 237.6]
  Anti-HPV 11: number analyzed (Participants) | 328
  Anti-HPV 11 | 172.1 [158.3 to 187.1]
  Anti-HPV 16: number analyzed (Participants) | 338
  Anti-HPV 16 | 1025.8 [945.5 to 1113.0]
  Anti-HPV 18: number analyzed (Participants) | 320
  Anti-HPV 18 | 228.0 [204.4 to 254.4]

13. Primary Outcome: Extension Stage: GMTs for Serum Anti-HPV Types 6, 11, 16, and 18 at Month 24 Assessed by Immunoglobulin G Luminex Immunoassay (IgG LIA)
Description: as for outcome 12
Time Frame: Month 24 post-vaccination 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Years
Number analyzed (Participants) | 365
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 322
  Anti-HPV 6 | 85.5 [76.4 to 95.6]
  Anti-HPV 11: number analyzed (Participants) | 322
  Anti-HPV 11 | 68.6 [61.6 to 76.4]
  Anti-HPV 16: number analyzed (Participants) | 333
  Anti-HPV 16 | 394.9 [354.6 to 439.9]
  Anti-HPV 18: number analyzed (Participants) | 316
  Anti-HPV 18 | 76.9 [67.0 to 88.3]

14. Primary Outcome: Extension Stage: GMTs for Serum Anti-HPV Types 6, 11, 16, and 18 at Month 36 Assessed by Immunoglobulin G Luminex Immunoassay (IgG LIA)
Description: as for outcome 12
Time Frame: Month 36 post-vaccination 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Years
Number analyzed (Participants) | 365
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 318
  Anti-HPV 6 | 66.5 [59.6 to 74.1]
  Anti-HPV 11: number analyzed (Participants) | 318
  Anti-HPV 11 | 52.7 [47.2 to 58.8]
  Anti-HPV 16: number analyzed (Participants) | 329
  Anti-HPV 16 | 304.0 [272.2 to 339.5]
  Anti-HPV 18: number analyzed (Participants) | 312
  Anti-HPV 18 | 57.5 [50.0 to 66.1]

15. Primary Outcome: Extension Stage: GMTs for Serum Anti-HPV Types 6, 11, 16, and 18 at Month 48 Assessed by Immunoglobulin G Luminex Immunoassay (IgG LIA)
Description: Serum antibody titers (Geometric mean titers) for HPV Types 6, 11, 16, and 18 were measured. Antibodies were measured using IgG LIA.
Time Frame: Month 48 post-vaccination 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Year
Number analyzed (Participants) | 365
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 311
  Anti-HPV 6 | 63.4 [56.8 to 70.8]
  Anti-HPV 11: number analyzed (Participants) | 311
  Anti-HPV 11 | 51.1 [45.9 to 56.9]
  Anti-HPV 16: number analyzed (Participants) | 321
  Anti-HPV 16 | 289.6 [258.7 to 324.2]
  Anti-HPV 18: number analyzed (Participants) | 305
  Anti-HPV 18 | 55.3 [47.8 to 63.9]

16. Primary Outcome: Extension Stage: GMTs for Serum Anti-HPV Types 6, 11, 16, and 18 at Month 60 Assessed by Immunoglobulin G Luminex Immunoassay (IgG LIA)
Description: as for outcome 15
Time Frame: Month 60 post-vaccination 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Year
Number analyzed (Participants) | 365
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 307
  Anti-HPV 6 | 58.6 [52.5 to 65.4]
  Anti-HPV 11: number analyzed (Participants) | 307
  Anti-HPV 11 | 47.2 [42.4 to 52.5]
  Anti-HPV 16: number analyzed (Participants) | 317
  Anti-HPV 16 | 264.3 [235.8 to 296.3]
  Anti-HPV 18: number analyzed (Participants) | 302
  Anti-HPV 18 | 51.0 [44.0 to 59.1]

17. Primary Outcome: Extension Stage: Percentage of Participants With Seropositivity to HPV Types 6, 11, 16, and 18 at Month 12 Assessed by IgG LIA
Description: The percentage of participants who are seropositive to each of HPV Types 6, 11, 16, and 18 were assessed. Antibodies were measured using IgG LIA.
Time Frame: Month 12 post-vaccination 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Year
Number analyzed (Participants) | 365
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 328
  Anti-HPV 6 | 100.0 [98.9 to 100.0]
  Anti-HPV 11: number analyzed (Participants) | 328
  Anti-HPV 11 | 100.0 [98.9 to 100.0]
  Anti-HPV 16: number analyzed (Participants) | 338
  Anti-HPV 16 | 100.0 [98.9 to 100.0]
  Anti-HPV 18: number analyzed (Participants) | 320
  Anti-HPV 18 | 100.0 [98.9 to 100.0]

18. Primary Outcome: Extension Stage: Percentage of Participants With Seropositivity to HPV Types 6, 11, 16, and 18 at Month 24 Assessed by IgG LIA
Description: as for outcome 17
Time Frame: Month 24 post-vaccination 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Year
Number analyzed (Participants) | 365
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 322
  Anti-HPV 6 | 98.4 [96.4 to 99.5]
  Anti-HPV 11: number analyzed (Participants) | 322
  Anti-HPV 11 | 98.4 [96.4 to 99.5]
  Anti-HPV 16: number analyzed (Participants) | 333
  Anti-HPV 16 | 100.0 [98.9 to 100.0]
  Anti-HPV 18: number analyzed (Participants) | 316
  Anti-HPV 18 | 98.1 [95.9 to 99.3]

19. Primary Outcome: Extension Stage: Percentage of Participants With Seropositivity to HPV Types 6, 11, 16, and 18 at Month 36 Assessed by IgG LIA
Description: as for outcome 17
Time Frame: Month 36 post-vaccination 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Year
Number analyzed (Participants) | 365
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 318
  Anti-HPV 6 | 98.1 [95.9 to 99.3]
  Anti-HPV 11: number analyzed (Participants) | 318
  Anti-HPV 11 | 99.4 [97.7 to 99.9]
  Anti-HPV 16: number analyzed (Participants) | 329
  Anti-HPV 16 | 100.0 [98.9 to 100.0]
  Anti-HPV 18: number analyzed (Participants) | 312
  Anti-HPV 18 | 96.2 [93.4 to 98.0]

20. Primary Outcome: Extension Stage: Percentage of Participants With Seropositivity to HPV Types 6, 11, 16, and 18 at Month 48 Assessed by IgG LIA
Description: as for outcome 17
Time Frame: Month 48 post-vaccination 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Year
Number analyzed (Participants) | 365
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 311
  Anti-HPV 6 | 97.4 [95.0 to 98.9]
  Anti-HPV 11: number analyzed (Participants) | 311
  Anti-HPV 11 | 98.4 [96.3 to 99.5]
  Anti-HPV 16: number analyzed (Participants) | 321
  Anti-HPV 16 | 100.0 [98.9 to 100.0]
  Anti-HPV 18: number analyzed (Participants) | 305
  Anti-HPV 18 | 95.1 [92.0 to 97.2]

21. Primary Outcome: Extension Stage: Percentage of Participants With Seropositivity to HPV Types 6, 11, 16, and 18 at Month 60 Assessed by IgG LIA
Description: as for outcome 17
Time Frame: Month 60 post-vaccination 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Year
Number analyzed (Participants) | 365
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 307
  Anti-HPV 6 | 96.7 [94.1 to 98.4]
  Anti-HPV 11: number analyzed (Participants) | 307
  Anti-HPV 11 | 98.4 [96.2 to 99.5]
  Anti-HPV 16: number analyzed (Participants) | 317
  Anti-HPV 16 | 100.0 [98.8 to 100.0]
  Anti-HPV 18: number analyzed (Participants) | 302
  Anti-HPV 18 | 95.4 [92.3 to 97.4]

22. Secondary Outcome: Base Stage: Percentage of Participants With Seroconversion for HPV Types 6, 11, 16, and 18: cLIA
Description: Seroconversion is defined as changing serostatus from seronegative at Day 1 to seropositive at 1 month post dose 3. Antibodies were measured using a Competitive Luminex Immunoassay (cLIA). Antibody titers were expressed as milli Merck Units/milliliter (mMU/mL).
Time Frame: Month 7 (1 month postdose 3)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Base Study: Chinese Girls Aged 9 to 19 Years | Base Study: Chinese Young Women Aged 20 to 26 Years
Number analyzed (Participants) | 383 | 383
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 343 | 315
  Anti-HPV 6 | 100.0 | 100.0
  Anti-HPV 11: number analyzed (Participants) | 343 | 315
  Anti-HPV 11 | 100.0 | 100.0
  Anti-HPV 16: number analyzed (Participants) | 354 | 330
  Anti-HPV 16 | 100.0 | 100.0
  Anti-HPV 18: number analyzed (Participants) | 333 | 318
  Anti-HPV 18 | 100.0 | 100.0
Statistical Analysis 1: Comparison: Base Study: Chinese Girls Aged 9 to 19 Years vs Base Study: Chinese Young Women Aged 20 to 26 Years; Difference of Seroconversion percentage HPV 6; Test type: Non-Inferiority — The statistical criterion for non-inferiority required that the lower bound of two-sided 95% confidence interval for the difference (9 to 19 years old minus 20 to 26 years old) in seroconversion percentages being greater than -5 percentage points for each HPV type; p < 0.0001, Miettinen & Nurminen method; Difference in percentages (%) = 0.0, 95% CI 2-sided [-1.1 to 1.2]
Statistical Analysis 2: Comparison: Base Study: Chinese Girls Aged 9 to 19 Years vs Base Study: Chinese Young Women Aged 20 to 26 Years; Difference of Seroconversion percentage HPV 11; Test type: Non-Inferiority — [test comment as in outcome 22, analysis 1]; p < 0.0001, Miettinen & Nurminen method; Difference in percentages (%) = 0.0, 95% CI 2-sided [-1.1 to 1.2]
Statistical Analysis 3: Comparison: Base Study: Chinese Girls Aged 9 to 19 Years vs Base Study: Chinese Young Women Aged 20 to 26 Years; Difference of Seroconversion percentage HPV 16; Test type: Non-Inferiority — [test comment as in outcome 22, analysis 1]; p < 0.0001, Miettinen & Nurminen method; Difference in percentages (%) = 0.0, 95% CI 2-sided [-1.1 to 1.2]
Statistical Analysis 4: Comparison: Base Study: Chinese Girls Aged 9 to 19 Years vs Base Study: Chinese Young Women Aged 20 to 26 Years; Difference of Seroconversion percentage HPV 18; Test type: Non-Inferiority — [test comment as in outcome 22, analysis 1]; p < 0.0001, Miettinen & Nurminen method; Difference in percentages (%) = 0.0, 95% CI 2-sided [-1.1 to 1.2]

23. Secondary Outcome: Base Stage: Geometric Mean Titers for Serum Anti-HPV Types 6, 11, 16, and 18: IgG LIA
Description: Antibodies to HPV Types 6, 11, 16, and 18 were measured using an IgG LIA. Antibody titers were expressed as milli Merck Units/milliliter (mMU/mL).
Time Frame: Month 7 (1 month postdose 3)
Population: All participants who received the correct dose of all 3 study vaccinations within visit window; was seronegative at Day 1 for the human papilloma virus (HPV) type being analyzed; provided Month 7 serum sample within visit window; and did not meet any exclusion criteria at any time during base stage.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Base Study: Chinese Girls Aged 9 to 19 Years | Base Study: Chinese Young Women Aged 20 to 26 Years
Number analyzed (Participants) | 383 | 383
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 343 | 315
  Anti-HPV 6 | 902.7 [831.2 to 980.3] | 604.5 [554.7 to 658.8]
  Anti-HPV 11: number analyzed (Participants) | 343 | 315
  Anti-HPV 11 | 756.2 [695.7 to 821.9] | 518.7 [475.5 to 565.9]
  Anti-HPV 16: number analyzed (Participants) | 354 | 330
  Anti-HPV 16 | 4170.0 [3849.3 to 4517.4] | 2659.3 [2447.8 to 2889.0]
  Anti-HPV 18: number analyzed (Participants) | 333 | 318
  Anti-HPV 18 | 1012.8 [918.7 to 1116.5] | 612.0 [553.9 to 676.1]

24. Secondary Outcome: Base Stage: Percentage of Participants With Seroconversion for HPV Types 6, 11, 16, and 18: IgG LIA
Description: The percentage of participants who seroconverted to each of HPV Types 6, 11, 16, and 18 was assessed. Antibodies were measured using IgG LIA.
Time Frame: Month 7 (1 month postdose 3)
Population: as for outcome 23
Measure: Number; unit: Percentage of Participants
Arm/Group | Base Study: Chinese Girls Aged 9 to 19 Years | Base Study: Chinese Young Women Aged 20 to 26 Years
Number analyzed (Participants) | 383 | 383
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 343 | 315
  Anti-HPV 6 | 100.0 | 100.0
  Anti-HPV 11: number analyzed (Participants) | 343 | 315
  Anti-HPV 11 | 100.0 | 100.0
  Anti-HPV 16: number analyzed (Participants) | 354 | 330
  Anti-HPV 16 | 100.0 | 100.0
  Anti-HPV 18: number analyzed (Participants) | 333 | 318
  Anti-HPV 18 | 100.0 | 100.0

25. Secondary Outcome: Base Stage: Percentage of Participants Who Experienced a Solicited Injection-site Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Solicited injection-site AEs included injection-site redness, swelling, induration, pain, and pruritus.
Time Frame: Up to 15 days after any vaccination
Population: The analysis population concisted of participants who recieved at least one dose of study vaccination.
Measure: Number; unit: Percentage of Participants
Arm/Group | Base Study: Chinese Girls Aged 9 to 19 Years | Base Study: Chinese Young Women Aged 20 to 26 Years
Number analyzed (Participants) | 383 | 383
Percentage of Participants | 36.6 | 40.7

26. Secondary Outcome: Base Stage: Percentage of Participants Participants Who Experienced a Solicited Systemic AE
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Solicited systemic AEs included hypersensitivity, headache, fatigue, vomiting, nausea, diarrhea, myalgia, pyrexia, and cough.
Time Frame: Up to 15 days after any vaccination
Population: The analysis population concisted of participants who recieved at least one dose of study vaccination.
Measure: Number; unit: Percentage of Participants
Arm/Group | Chinese Girls Aged 9 to 19 Years | Base Study: Chinese Young Women Aged 20 to 26 Years
Number analyzed (Participants) | 383 | 383
Percentage of Participants | 39.9 | 42.0

27. Secondary Outcome: Base Stage: Percentage of Participants Who Experienced a Serious Adverse Event (SAE)
Description: An SAE is an AE that results in death, is life threatening, requires hospitalization or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, according to medical or scientific judgment, may jeopardize the participant or requires medical or surgical intervention to prevent one of the other outcomes listed in the above definition.
Time Frame: Up to Month 7 (1 month postdose 3)
Population: The analysis population concisted of participants who recieved at least one dose of study vaccination.
Measure: Number; unit: Percentage of Participants
Arm/Group | Chinese Girls Aged 9 to 19 Years | Base Study: Chinese Young Women Aged 20 to 26 Years
Number analyzed (Participants) | 383 | 383
Percentage of Participants | 1.6 | 2.87

28. Secondary Outcome: Base Stage: Percentage of Participants Who Experienced an AE
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment
Time Frame: Up to 31 days after any vaccination
Population: The analysis population concisted of participants who recieved at least one dose of study vaccination.
Measure: Number; unit: Percentage of Participants
Arm/Group | Chinese Girls Aged 9 to 19 Years | Base Study: Chinese Young Women Aged 20 to 26 Years
Number analyzed (Participants) | 383 | 383
Percentage of Participants | 61.6 | 68.9

29. Secondary Outcome: Base Stage: Maximum Axillary Temperature: Merck Sharp & Dohme (MSD) Criteria
Description: In the global studies, fever is defined as an oral temperature of ≥37.8°C or 100.0°F, which is equivalent to axillary temperature of ≥37.2°C, while the definition of fever is axillary temperature of ≥37.1°C in Chinese criteria. To be compliant to Chinese criteria, axillary temperatures of ≥37.1°C was considered as a fever in this study. Body temperature readings assessed orally were converted to the axillary equivalent. The percentage of participants with a maximum axillary or converted axillary temperature was summarized by temperature range.
Time Frame: Up to 5 days after any vaccination
Population: The analysis population concisted of participants who recieved at least one dose of study vaccination.
Measure: Number; unit: Percentage of Participants
Arm/Group | Chinese Girls Aged 9 to 19 Years | Base Study: Chinese Young Women Aged 20 to 26 Years
Number analyzed (Participants) | 383 | 383
Percentage of Participants
  < 37.2 °C (99.0 °F) | 87.2 | 84.9
  ≥37.2 °C (99.0 °F) and < 38.3 °C (100.9 °F) | 12.3 | 14.9
  ≥ 38.3 °C (100.9 °F) and < 39.3 °C (102.7 °F) | 0.3 | 0.3
  ≥ 39.3 °C (102.7 °F) and < 40.3 °C (104.5 °F) | 0.3 | 0.0
  ≥ 40.3 °C (104.5 °F) | 0.0 | 0.0

30. Secondary Outcome: Extension Stage: Percentage of Participants Who Experienced an SAE
Description: The percentage of participants with an SAE will be assessed. An SAE is an AE that results in death, is life threatening, requires hospitalization or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, according to medical or scientific judgment, may jeopardize the participant or requires medical or surgical intervention to prevent one of the other outcomes listed in the above definition.
Time Frame: Month 7 up to Month 60
Population: The analysis population consisted of all participants who received at least 1 dose of study vaccination and had clinical follow-up for safety.
Measure: Number; unit: Percentage of Participants
Arm/Group | Extension Study: Chinese Girls Aged 9 to 19 Years
Number analyzed (Participants) | 365
Percentage of Participants | 2.2

ADVERSE EVENTS:
Time Frame: Base Stage only: Up to approximately 7 months Extension Stage: Month 7 up to approximately 60 Months
Description: All participants who received at least 1 vaccination.
Arm/Group | Base Study: Chinese Girls Aged 9 to 19 Years | Base Study: Chinese Young Women Aged 20 to 26 Years | Extension Study: Chinese Girls Aged 9 to 19 Years
All-Cause Mortality (participants affected / at risk) | 0/383 | 0/383 | 0/365
Serious Adverse Events (participants affected / at risk) | 6/383 | 11/383 | 8/365
Other Adverse Events (participants affected / at risk) | 216/383 | 238/383 | 0/365
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Study: Chinese Girls Aged 9 to 19 Years (N=383) | Base Study: Chinese Young Women Aged 20 to 26 Years (N=383) | Extension Study: Chinese Girls Aged 9 to 19 Years (N=365)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Hypertrophic anal papilla (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bacterial vulvovaginitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Complicated appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Peroneal nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Sciatic nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (2)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal somatic symptom disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus urethral (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrosalpinx (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Mammary duct ectasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic adhesions (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vulval eczema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Study: Chinese Girls Aged 9 to 19 Years (N=383) | Base Study: Chinese Young Women Aged 20 to 26 Years (N=383) | Extension Study: Chinese Girls Aged 9 to 19 Years (N=365)
Diarrhoea (Gastrointestinal disorders) | 15 (18) | 31 (33) | 0 (0)
Fatigue (General disorders) | 41 (59) | 42 (57) | 0 (0)
Injection site pain (General disorders) | 122 (189) | 152 (233) | 0 (0)
Injection site pruritus (General disorders) | 32 (33) | 16 (20) | 0 (0)
Injection site swelling (General disorders) | 22 (25) | 11 (14) | 0 (0)
Pyrexia (General disorders) | 104 (196) | 108 (194) | 0 (0)
Headache (Nervous system disorders) | 32 (47) | 42 (51) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 37 (40) | 41 (47) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 29 (30) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the sponsor, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission. This allows the sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT03493542/Prot_SAP_001.pdf